CLINICAL TRIAL: NCT05868122
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Multidose Clinical Trial to Evaluate a Fixed Combination of Acetaminophen/Naproxen Sodium in Acute Postoperative Pain Following Bunionectomy
Brief Title: A Study to Evaluate a Fixed Combination of Acetaminophen/Naproxen Sodium in Acute Postoperative Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCSPAA005197; CCSPAA005197 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acetaminophen/Naproxen Sodium Fixed Combination (Experimental): Participants will receive oral doses of two Acetaminophen/Naproxen Sodium Fixed Combination tablets taken with water. Multiple doses will be administered over a 48-hour period.
  Interventions: Drug: Acetaminophen/Naproxen Sodium Fixed Combination
- Placebo (Placebo Comparator): Participants will receive oral doses of two placebo tablets taken with water. Multiple doses will be administered over a 48-hour period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen/Naproxen Sodium Fixed Combination — Fixed combination of Acetaminophen/Naproxen Sodium will be administered orally.
  Arms: Acetaminophen/Naproxen Sodium Fixed Combination
Drug: Placebo — Placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate effectiveness of a fixed combination of acetaminophen/naproxen sodium compared with placebo for reduction of pain when administered as multiple doses over a 48-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Females have a negative urine pregnancy at screening and on the morning of surgery
* Weight of 100 pounds or greater and have a body mass index (BMI) of 17.5 to 38.0 (inclusive) at screening
* Scheduled to undergo primary, unilateral, distal, first metatarsal bunionectomy (osteotomy and internal fixation) with no additional collateral procedures. Participants who have previously undergone bunionectomy on the contralateral foot will not be prohibited from enrolling in this study if performed greater than or equal to (>=) 6 months
* Are able to comprehend and follow the requirements of the study (including pre-surgical instructions provided by the site and availability on scheduled visit dates) based upon research site personnel's assessment
* Provide written informed consent (for participants who are below the age of legal consent, parent or legally authorized representative provides written informed consent and the participant provides written assent)
* Participant agrees to the contraceptive requirements
* Are willing for this to be the only investigational product used during the study
* Have a negative urine drug screen at screening, and on day of surgical procedure. a) a positive drug screen for a known prescribed concomitant medication that is not otherwise exclusionary will not disqualify a participant; b) drug and alcohol screen results must be negative for a participant to receive study medication, a positive Tetrahydrocannabinol (THC) screen will only be exclusionary on day of surgery (Day 0)

Postoperative Inclusion Criteria

* Participant reports both of the following after discontinuation of the popliteal block and before 2:00 PM on Day 1. a) moderate or severe pain on a 4-point categorical pain rating scale (with categories of none, mild, moderate, or severe; b) a score >= 5 on 11-point pain intensity-numerical pain rating scale (PI-NRS)
* Participant is able to answer questions and follow commands, and appropriately participate in requisite pain evaluation assessments dictated in the protocol
* The surgical procedure from incision to closure was not longer than 2 hours
* The participant has had no evidence of respiratory insufficiency, clinically significant hypotension, brady cardia, or any other abnormality, during or following surgery that, in the Investigator's opinion, significantly increases the risks of study drug administration
* There were no significant deviations from the surgical protocol, anesthetic protocol, or specified analgesic regimen, that would, in the opinion of the Investigator, put the participant at risk of participation in the trial, confound the analgesic endpoints of the trial or cause concern regarding the participants ability to participate in the trial

Exclusion Criteria:

* Are female and are pregnant, breastfeeding, or currently trying to become pregnant
* Are male with a pregnant partner or a partner who is currently trying to become pregnant
* Have a known allergy or hypersensitivity to: a) naproxen or other nonsteroidal anti-inflammatory drugs, including aspirin; b) oxycodone or other opioids; c) acetaminophen; d) any other drug listed in the surgical and anesthetic protocol or postoperative pain management of the study protocol
* Have presence or a history of major medical condition that in the investigator's opinion may jeopardize the participant's safety or well-being, or the integrity of the study, example; a) hepatic, renal, pancreatic, gastrointestinal, cardiovascular, cerebrovascular, or thyroid diseases; b) history of head injury or seizures; c) history of respiratory depression or lung problems such as but not limited to asthma or chronic obstructive pulmonary disease; d) psychiatric disorders (although participants with well-controlled depression or anxiety, who are on a stable dose of medication may be allowed); e) problems urinating; f) history of blockage or narrowing of the stomach or intestines; g) uncontrolled hypertension indicated as systolic blood pressure >=160 millimetres of mercury (mmHg) or diastolic blood pressure >=100 mmHg. Blood pressure may be repeated after the participant has remained in a rested state for at least 10 minutes. The final blood pressure value will be used for eligibility; h) uncontrolled diabetes, as determined by the investigator, in the last six months; i) medical conditions that would interfere with normal pain perception (example diabetic neuropathy) in the opinion of the Investigator
* Have a history of endoscopically documented peptic ulcer disease or bleeding disorder in the last two years
* Are not able to swallow whole large tablets or capsules
* Participants will be excluded from the study for any of the following:a) routine use of oral analgesics >=3 times per week for a medical condition unrelated to bunion pain in the 2 months prior to surgery; b) opioid tolerant, that is, the participant is currently taking or has taken a chronic opioid for pain at a dose greater than or equal to 10 milligrams (mg) hydrocodone per day, more than 1 out of 7 days per week, in the 2 months prior to surgery; c. History of chronic tranquilizer use, heavy drinking, opioid abuse, or other substance abuse, as judged by the Investigator, in the last five years. Heavy drinking is defined as the use of more than four standard drinks daily or more than 14 drinks a week for men, and more than three standard drinks daily or more than seven standard drinks in a week for women. Standard drink refers to 14 grams (g) (0.6 ounce [oz.]) of pure alcohol, which is approximately 12 oz. of beer, 8 oz. of malt liquor, 5 oz. of wine, 1.5 oz. or "shot" of 80 proof distilled spirits or liquor (example., gin, rum, vodka, or whiskey); d) use of any immunosuppressive drugs, corticosteroids (except for topical corticosteroids), or injectable or oral anticoagulants (example., heparin, Lovenox, Xarelto, Eliquis, Pradaxa, Coumadin, Miradon) within 2 weeks prior to surgery; e) use of monoamine oxidase inhibitors within 2 weeks prior to surgery; f) use of alcohol within 24 hours prior to surgery; g) consumption of methylxanthine containing products (example, chocolate bars or chocolate beverages, coffee, tea, cola or caffeinated energy drinks), tobacco, or nicotine containing products (example, cigarettes, cigars, nicotine replacement therapies, vaping devices) less than (<) 12 hours prior to surgery; h) use of any other over-the-counter or prescription medications or supplements that, in the Investigator's opinion, may cause participation in the study to jeopardize the participant's safety or well-being, or may jeopardize the integrity of the study, within 5 days (or longer if the investigator deems a longer washout is warranted) prior to surgery
* Have a positive test for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV)
* Have participated in any interventional clinical trials within 30 days before screening
* Are related to those persons involved directly or indirectly with the conduct of this study (that is., Principal Investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson [J&J] subsidiaries, contractors of J&J, and the families of each)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Time-weighted Sum of Pain Intensity Difference Score from 0 to 24 Hours After Dosing (SPID 0-24) | 0 to 24 hours post-dose
  Time-weighted SPID scores will be calculated using values collected on the Pain Intensity-Numerical Rating Scale (PI-NRS) ranging from 0-10 (0 = no pain, 10 = very severe pain) collected at each scheduled timepoint within the specified timeframe.

SECONDARY OUTCOMES:
Time-weighted SPID Score from 0 to 12 Hours After Dosing (SPID 0-12) | 0-12 hours post-dose
  Time-weighted SPID scores will be calculated using values collected on the PI-NRS ranging from 0-10 (0 = no pain, 10 = very severe pain) collected at each scheduled timepoint within the specified timeframe.
Time-weighted SPID from 0 to 48 Hours After Dosing (SPID 0-48) | 0-48 hours post-dose
  Time-weighted SPID scores will be calculated using values collected on PI-NRS ranging from 0-10 (0 = no pain, 10 = very severe pain) collected at each scheduled timepoint within the specified timeframe.
Time to Confirmed Perceptible Pain Relief (TCPR) | Up to 12 hours
  TCPR is defined as the time (in minutes) to perceptible pain relief as indicated on the first stopwatch, provided that the participant also stopped the second stopwatch indicating meaningful pain relief.
Time to Meaningful Pain Relief (TMPR) | Up to 12 hours
  TMPR is defined as the time (in minutes) to meaningful pain relief as indicated on the second stopwatch.
Time to First use of Rescue Medication | Up to 48 hours
  Time to first use of rescue medication will be measured as the elapsed time from when investigational product was given until the time rescue medication was first given.
Percentage of Participants who use Rescue Medication During the First 12 Hours | Up to 12 hours
  Percentage of participants who use rescue medication during the first 12 hours will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Consumer Inc. (J&JCI) Clinical Trial, Study Director — Johnson & Johnson Consumer Inc. (J&JCI)
Locations (4):
- United States (4):
  - Lotus Clinical Research, LLC, New Providence, New Jersey
  - First Surgical Hospital, Bellaire, Texas
  - The Heights Hospital / Memorial Herman Village, Houston, Texas
  - Endeavor Clinical Trails, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu